CLINICAL TRIAL: NCT05642286
Title: Prospective, Multi Center, Single Group Target Value Study to Evaluate the Safety and Effectiveness of Endovascular Interventional Device Control System and Supporting Consumables for Coronary Intervention
Brief Title: Clinical Study of Endovascular Interventional Surgical Instrument Control System and Related Consumables in Percutaneous Coronary Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Operation Robot Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMLY3001-01A
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-10

CONDITIONS: Percutaneous Coronary Intervention; Coronary Heart Disease; Robotic Surgical Procedures
Keywords: Robotic Surgical Procedures; PCI; CHD
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Intervention Model Description: prospective, multi center, single group target value design is adopted; 218 subjects who met the inclusion criteria and did not meet the exclusion criteria were planned to be included in the study, and the trial medical devices were used to assist surgery and complete follow-up, so as to evaluate the safety and effectiveness of the trial medical devices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot assisted surgery group (Experimental): robotic-assisted PCI
  Interventions: Device: ALLVAS® robotic-assisted PCI

INTERVENTIONS:
Device: ALLVAS® robotic-assisted PCI — ALLVAS® robotic-assisted PCI

SUMMARY:
The goal of this study is to evaluate the safety and effectiveness of endovascular interventional surgery instrument control system （ALLVAS®robot）and supporting consumables for coronary artery interventional surgery.

Participants will will complete coronary intervention surgery with the assistance of robot system（ALLVAS®robot）, and evaluate the effect of the use effect of robots and clinical treatment after surgery

DETAILED DESCRIPTION:
Interventional therapy plays an important role in the treatment of coronary heart disease. At present, the main treatment methods still rely on human hands, and there are some defects, including but not limited to hand shaking and visual error. The use of robots may partly circumvent the above shortcomings.

This study is to evaluate the safety and effectiveness of ALLVAS®robot for coronary artery interventional surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily participate in and sign the informed consent form, and can cooperate to complete the whole trial process;
2. aged over 18 and under 75;
3. After coronary CT angiography (CTA) or coronary angiography (DSA), the investigator judged that the patients who needed interventional blood supply reconstruction (target vessel diameter ≥ 2.5mm and lesion stenosis ≥ 70%).

Exclusion Criteria:

1. Acute myocardial infarction occurred within 7 days;
2. The target vessel has received coronary intervention within 30 days;
3. Restenosis in stent of target vessel;
4. Patients with bifurcation lesions whose target vessel branches need to be protected but cannot protect the collateral branches;
5. Hemodynamic instability (including low blood pressure or use of vasopressors to maintain blood pressure;)
6. Three vessel lesions;
7. The target vessel was diagnosed as coronary chronic occlusive disease (CTO) or left main artery stenosis or severe calcification requiring pretreatment;
8. Perforation, dissection or aneurysm of the proximal vessel of the target vessel;
9. Echocardiography showed that left ventricular ejection fraction (LVEF) was less than 50%;
10. Stroke or transient ischemic attack (TIA) occurred within 30 days;
11. Peptic ulcer or gastrointestinal bleeding within 90 days;
12. Estimated glomerular filtration rate eGFR (ckd epi)<30 ml/min/1.73 m2;
13. Platelet count<50 × 109/L or > 700 × 109/L； White blood cell count < 3 × 109/L;
14. Women who are in pregnancy or lactation or have a pregnancy preparation plan during the trial period;
15. People with allergy history or contraindication to antiplatelet drugs, anticoagulants, anesthetics, contrast agents, stent materials and their coating drugs;
16. Severe infections difficult to control;
17. Those who have mental diseases or mental disorders and cannot be described normally;
18. Emergency operation is required for any reason;
19. Those who have participated in clinical trials of other drugs or medical devices within 3 months before screening;
20. The investigator believes that there are other circumstances that are not suitable for this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients With Device Technical Success | 1 day
  Defined as after the operator completed intracoronary therapy of coronary artery with robot assistance, the ratio of successful subjects with instrument technology among all enrolled subjects was reached.
Percentage of Participants With Clinical Procedural Success | 3 days or hospital discharge, whichever occurs first
  Defined as after the operator completed intracoronary coronary artery therapy with robot assistance, the ratio of clinically successful subjects among all enrolled subjects was reached.

SECONDARY OUTCOMES:
The Ratio Between the Radiation Exposure of the Primary Operator and the Radiation Exposure at the Table | 1 day
  Defined as the difference between the radiation exposure measured at the procedure table (the conventional site of the primary operator) and the radiation exposure measured at the primary operator's position during the procedure.
Evaluation of operational performance of experimental medical devices | 1 day
  Multiple evaluation forms, including those for stability, operation convenience,interface friendliness, image clarity, need to be completed postoperatively by operator. These include one or more levels such as excellent, good, general, poor, etc.
  Stability refers to whether the operator has any abnormal situation during the use of the device; Operation convenience refers to whether the operator is smooth in the process of using the instrument.
  Interface friendliness and image clarity refer to whether the operator has any doubt or confusion about the interface image feedback during the use of the instrument and the clarity of the interface image during operation.